CLINICAL TRIAL: NCT01071031
Title: A Multicentre, Two Stage, Randomised, Double Blind Study of the Safety, Tolerability and Immunogenicity of a Human Immunodeficiency Virus (HIV) Vaccine Candidate, HIV-v
Brief Title: HIV Vaccine Study in HIV Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepTcell Limited (Industry)
Responsible Party: Dr. Stuart Robinson, Head of Business Development, PepTcell Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HIV-v-001
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Safety; Tolerability; Immunogenicity; Human Immunodeficiency Virus; HIV-1; Vaccine; CD4; Viral Load; HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Low Dose HIV-v with water for injection
  Interventions: Biological: HIV-v (Low Dose)
- Group 2 (Experimental): Low Dose HIV-v with adjuvant
  Interventions: Biological: HIV-v (Low Dose)
- Group 3 (Experimental): High Dose HIV-v with water for injection
  Interventions: Biological: HIV-v (High Dose)
- Group 4 (Experimental): High Dose HIV-v with adjuvant
  Interventions: Biological: HIV-v (High Dose)
- Group 5 (Placebo Comparator): Control group: adjuvant only or water for injection only
  Interventions: Biological: HIV-v (Control)

INTERVENTIONS:
Biological: HIV-v (Low Dose) — Low Dose HIV-v (a sterile lyophilised mixture of polypeptide T-cell epitope sequences) with water for injection or adjuvant
  Administration: A single subcutaneous injection
  Arms: Group 1; Group 2
Biological: HIV-v (High Dose) — High Dose HIV-v (a sterile lyophilised mixture of polypeptide T-cell epitope sequences with water for injection or adjuvant
  Administration: A single subcutaneous injection
  Arms: Group 3; Group 4
Biological: HIV-v (Control) — Adjuvant only or Water for injection only
  Administration: A single subcutaneous injection
  Arms: Group 5

SUMMARY:
The purpose of the study is to see whether a single vaccination (injection) with the investigational HIV vaccine is safe and effective in patients who are HIV positive but have not yet begun anti-retroviral therapy. As this is an exploratory study, four different dose formulations of HIV vaccine will be investigated.

This study will evaluate whether or not the HIV vaccine is able to reduce the HIV viral load (number of HIV virus particles in the blood) and increase or slow the decline in CD4 T cell count.

DETAILED DESCRIPTION:
The study will consist of a screening period of 3 to 21 days before vaccination on Day 0 and a double-blind treatment period of 28 days with a follow up period of 5 months. Prior to conducting any study-related procedures, subjects will provide written informed consent. During screening, eligibility will be assessed, a medical history will be taken, a complete physical examination will be performed and vital signs will be measured. Blood samples will be taken for the assessment of HCV and HBV status. Further samples will be taken for CD4 and HIV load, haematology, biochemistry, urinalysis and a 12-lead electrocardiographic (ECG) assessment will be carried out. A self-assessment diary card will be used by subjects between Day 0 and Day 28 to record any AEs.

On Days 7, 14, 21 and 28 an AE interview will be conducted, concomitant medications and vital signs will be recorded and a physical examination will be performed. Samples will be collected for haematology, clinical chemistry and urinalysis. In addition, samples will be collected for CD4 T cell count and HIV viral load at days 14 and 28 after vaccination. A sample will be collected for immunogenicity on Day 28.

All patients will attend follow-up visits at Weeks 8, 12, 16, 20 and 24 at which a physical examination and examination of the injection site will be performed and vital signs measured. Samples will be collected for haematology, biochemistry, urinalysis CD4 T-cell count and HIV viral load. Blood samples for immunogenicity testing will be collected at Weeks 12 and 24.

Stage I: Sequential, non-randomised, single blind, parallel group. Five male HIV-1 positive volunteers will be vaccinated in a sequential, non-randomised single blind fashion. They will each receive one of the five possible active study treatments (WFI only, adjuvant only, low dose + WFI, low dose + adjuvant, high dose + WFI and high dose + adjuvant). Each of these five patients will be observed as in-patients for 24 hours after vaccination and vaccinations will be performed in a sequential manner with at least 48 hours observation of each patient before vaccination of the next patient is commenced.

Following completion of the '28 day treatment follow up' by the five Stage I subjects a Safety Committee will review the safety and tolerability data for these subjects and will make a recommendation for continuing or discontinuing recruitment and any changes that may be required in the conduct of the study. Subject to a positive decision from the Safety Committee the remaining subjects will be recruited into Stage II of the study.

Stage II: randomised, double-blind group 50 male HIV-1 positive volunteers will be randomised to one of five possible treatment groups. Following completion of the Day 1 Visit by the first five subjects in Stage II the Safety Committee will review the blinded safety and tolerability data for these subjects. Subject to acceptable safety and tolerability, the centres will be allowed to continue recruitment for the rest of the planned cohort.

After 25 Stage II subjects have completed the Day 1 Visit a Safety Committee will review the blinded data generated and will make a recommendation for continuing or discontinuing recruitment and any changes that may be required in the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects age 18 - 50 years inclusive with HIV-1 infection
* Documented as HIV positive, with viral loads higher than 5,000 copies per millilitre of blood, but less than 500,000 using either a branched DNA test, or an RT-PCR test
* CD4 T cell count >350/mm3
* Clinically stable in the opinion of the investigator and not expected to require anti-retroviral therapy during the course of the study
* No evidence of any AIDS defining illness
* Subjects with male or female partners must agree to use a barrier method of protection against disease transmission during intercourse (e.g. condom).
* Subjects whose female partners are of child-bearing potential must also agree to use a second contraceptive method (e.g. spermicidal agent, IUD, hormonal contraceptive) in addition to a condom for the duration of the study.
* Provide written informed consent to participate in the study and be willing to comply with all study procedures.

Exclusion Criteria:

* Participation in a clinical trial or receipt of an experimental therapy within 30 days prior to study dosing
* Receipt of another vaccine 30 days before or 30 days after HIV-v
* Currently receiving anti-viral, anti-retroviral therapy or any chronic anti-infective therapy
* Receiving, or have received over the previous two weeks, any treatment that might modulate the immune response after vaccination, including, but not limited to, immunosuppressive therapy and systemic corticosteroids
* Suffers from a disease or is undergoing treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800µg/day beclometasone or equivalent), radiation treatment or cytotoxic drugs
* Received a blood transfusion or immunoglobulins within 90 days prior to study entry
* Patients on inhaled corticosteroids for asthma or other respiratory conditions
* Subjects having an infective exacerbation during the screening process as defined as a requirement of inhaled, oral, or intravenous antibiotics prior to the first study dose will be excluded
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) or any over-the-counter product, herbal product, diet aid, hormone supplement, etc., within 14 days prior to vaccination or any planned administration of these products over the course of the first 28 days after vaccination (unless approved by both the Principal Investigator and the Sponsor)
* Patients with Hepatitis B or C co-infection (though serological evidence of previous hepatitis C infection with no evidence of carrier status is acceptable)
* Suffers from or has a history of significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, haematological or renal disorder
* Subjects with clinically significant out of range laboratory values as stated in Section 8.6 of the protocol
* Patients with a history of significant or allergic reaction to vaccines
* Patients with a known or suspected dependence on illicit drugs or alcohol and those undergoing illicit drug replacement programmes
* Is direct employee of the study site or monitoring CRO

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety and tolerability of the PepTcell HIV vaccine by analysis of safety data including changes in HIV load and CD4 T cell count. | Pre-vaccination, days 1, 2, 7, 14, 21 and 28 after vaccination and weeks 8, 12, 16, 20 and 24 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD, Principal Investigator — St Stephen's Aids Trust; Stuart Robinson, Study Director — PepTcell Limited
Locations (5):
- United Kingdom (5):
  - Grahame Hayton Unit, Ambrose King Centre, Royal London Hospital, London, London
  - St. Stephen's Centre, Chelsea and Westminster Foundation Trust, London, London
  - Elton John Centre, Sussex House,, Brighton
  - North Manchester General Hospital, Department for Infectious Diseases, Manchester
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Boffito M, Fox J, Bowman C, Fisher M, Orkin C, Wilkins E, Jackson A, Pleguezuelos O, Robinson S, Stoloff GA, Caparros-Wanderley W. Safety, immunogenicity and efficacy assessment of HIV immunotherapy in a multi-centre, double-blind, randomised, Placebo-controlled Phase Ib human trial. Vaccine. 2013 Nov 19;31(48):5680-6. doi: 10.1016/j.vaccine.2013.09.057. Epub 2013 Oct 8. PMID 24120550